CLINICAL TRIAL: NCT02239068
Title: Residual Gastric Fluid With Administering Clear Liquids Within Two Hours of Anesthesia in Children
Brief Title: CT Residual Gastric Fluid Volume
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-0286
Record Dates: First submitted 2014-07-22; First posted 2014-09-12 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Clinical CT Abdomen/Pelvic With Oral Contrast and Sedation
Keywords: CT, sedation, oral contrast

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: The investigators hypothesize that more than 50% of the patients receiving enteric contrast material (ECM) < 2 hours of anesthesia/sedation would have residual gastric fluid volume (GFV) > 0.4 ml/kg. The investigators also hypothesize that measuring GFV by using region of interest in the CT technique is accurate compared to blind aspiration of the gastric contents with a syringe and a multi-orificed orogastric tube.

DETAILED DESCRIPTION:
The purpose of our study is to examine the residual gastric fluid volume when oral contrast is administered within 2 hours of anesthesia /sedation and to validate the accuracy of measuring the residual gastric volume by using region of interest in the CT image by using blind aspiration of the gastric contents with a syringe and a multi-orificed orogastric tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for CT abdomen with contrast and require anesthesia/sedation
* Subjects must be 1 month to 10 years of age (inclusive)
* The subject's legally authorized representative has given written informed consent to participate in the study

Exclusion Criteria:

* Subjects violate the institution fasting guideline before anesthesia /sedation with the exception of the oral contrast

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be recruited from the Radiology CT schedule.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Residual gastric fluid volume (GFV) < 0.4ml/kg or > 0.4 ml/kg | Approximately 2 hours
  Patients will have gastric volume suctioned and measured after the CT scan. The investigator will compare the amount suctioned to the measurement from the actual CT scan when all patients have been enrolled in the study.

SECONDARY OUTCOMES:
Residual gastric fluid volume (GFV) < 0.8 ml/kg or > 0.8 ml/kg | Approximate 2 hours
  Patients will have gastric volume suctioned and measured after the CT scan. The investigator will compare the amount suctioned to the measurement from the actual CT scan when all patients have been enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No